CLINICAL TRIAL: NCT05722782
Title: The Investigation of the Efficacity and Safety of Oral Non Steroidal Anti Inflammatory (NSAI) Drugs Such as Piroxicam as a Second Line Treatment of Patients Consulting the Emergency Department for Renal Colics
Brief Title: Oral NSAI Versus Acetaminophen or Placebo as a Discharge Treatment of Non Complicated Renal Colics
Acronym: NAP-RC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAP in RC
Record Dates: First submitted 2023-01-20; First posted 2023-02-10 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Renal Colic
Keywords: Renal Colic; NSAI; Acetaminophen
MeSH Terms: conditions — Renal Colic | interventions — Piroxicam; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NSAI (Active Comparator): Piroxicam: 20 mg per pill; one pill per day for five days
  Interventions: Drug: Piroxicam
- Acetaminophen (Active Comparator): Paracetamol: 1000 mg per day for five days
  Interventions: Drug: Acetaminophen
- Placebo (Placebo Comparator): Placebo: one pill per day for five days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Piroxicam — Patients allocated to this arm received , as a second line treatment of renal colics , a five days treatment with 20 mg piroxicam per day and were contacted at the seventh day by telephone call to investigate the efficacy and the side effects of the treatment
  Other Names: Piroxen
  Arms: NSAI
Drug: Acetaminophen — Patients allocated to this arm received , as a second line treatment of renal colics , a five days treatment with 1000 mg Acetaminophen per day and were contacted at the seventh day by telephone call to investigate the efficacy and the side effects of the treatment
  Arms: Acetaminophen
Drug: Placebo — Patients allocated to this arm received , as a second line treatment of renal colics , a five days treatment with placebo per day and were contacted at the seventh day by telephone call to investigate the efficacy and the side effects of the treatment
  Arms: Placebo

SUMMARY:
Treatment with NSAI in renal colics has not been well investigated and there is no clear recommendations regarding this subject.

The aim of this study is to determine if an oral NSAI treatment is beneficial in patients discharged for the emergency department after the first line treatment of a renal colic investigating the reccurence of pain, the reconsultation rates and the admissions.

DETAILED DESCRIPTION:
Renal colic (RC) are a frequent cause of consultation in the emergency departement (ED). It counts for approximatively 20 % of patients presenting to the ED with severe acute onset abdominal pain.

The first line treatment of renal colics is based on NSAI drugs associated with antalgics and is further investigated in the NSAI vs Morphine study (NCT02156596) But there is no clear recommendations regarding the outpatient treatment of renal colics. Oral NSAI are still widely used as a second line medicine for this condition and variety of molecules were tried with non solid scientific arguments.

Piroxicam, a non-selective COX inhibitor drug appared to the oxicam class of NSAI, is widely used to treat rhumatoid and inflammatory disesases, and often prescribed in Tunisia as a second line treatment of RC.

In this study, the investigators aimed to investigate the efficiency and safety of the use of oral NSAI drugs (piroxicam) compared to Acetaminophen or placebo as a second line treatment of renal colics

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Consenting to participate in the study
* Patients treated in the ED for RC
* No contraindications of NSAI or paracetamol treatment

Exclusion Criteria:

* Contraindication of NSAI treatment
* Patients non reachable by telephone call
* Patients that did not receive or use the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Efficacity of oral NSAI | 07 days
  The efficacity of the oral NSAI treatment was evaluated at the seventh day by a telephone call, asking for the reccurence of pain, the reconsultation rates and intervals and the need for other treatments (antalgics...)

SECONDARY OUTCOMES:
Safety of NSAI | 07 days
  Safety was evaluated by a telephone call asking for the occurence of NSAI side effects such as abdominal pain , vomiting , rush, bleeding or others

CONTACTS AND LOCATIONS:
Locations (1):
- Fattouma Bourguiba University Hospital, Monastir, Tunisia